CLINICAL TRIAL: NCT05542992
Title: Deep Learning Model Supplementary PET-CT as a More Effectively Diagnostic Method for Pure Solid Nodules Classification: a Multicenter Observational Study
Brief Title: Deep Learning Model for Pure Solid Nodules Classification
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Chen (Other)
Collaborators: Ningbo No.2 Hospital (Other); Zunyi Medical College (Other); The First Affiliated Hospital of Nanchang University (Other); The First Hospital of Lanzhou University, Gansu, China (Unknown)
Responsible Party: Sponsor-Investigator, Chang Chen, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Other Study IDs: L21-022
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Lung Cancer
Keywords: deep learning model; pure-solid nodules; PET-CT
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT-based deep learning model — CT-based deep learning model for pure-solid nodules classifications

SUMMARY:
The purpose of this study is to compare the predictive performance of a CT-based deep learning model for pure-solid nodules classification and compared with the tumor maximum standardized uptake value on PET in a multicenter prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Participants scheduled for surgery for radiological finding of pulmonary pure-solid lesions from the preoperative thin-section CT scans;
* The maximum short-axis diameter of lymph nodes less than 3 cm on CT scan;
* Age ranging from 18-75 years;
* definied pathological examination report available;
* Obtained written informed consent.

Exclusion Criteria:

* Multiple lung lesions;
* Poor quality of CT images;
* Participants with incomplete clinical information;
* Participants who have received neoadjuvant therapy before initial CT evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary radiological pure-solid nodules with size less than 3cm
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
AUC | 2022.01-2023.12
  Area under the curve of the receiver operating characteristic

SECONDARY OUTCOMES:
Accuracy | 2022.01-2023.12
  Ratio of the number of correctly classified samples to the total number of samples
sensitivity | 2022.01-2023.12
  The probability of detecting a positive test in the population with the gold standard for disease (positive)
Specificity | 2022.01-2023.12
  Odds of detecting a negative test in a population judged disease-free (negative) by the gold standard
PPV | 2022.01-2023.12
  Positive predictive value
NPV | 2022.01-2023.12
  Negative predictive value

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Shanghai Pulmonary Hospital, Yangpu, Shanghai Municipality
  - Lanzhou, China, Gansu
  - Zunyi, China, Guizhou
  - Nanchang, China, Jiangxi
  - Ningbo, China, Zhejiang

IPD SHARING:
Plan to Share IPD: No